CLINICAL TRIAL: NCT05848596
Title: The Effect of Simulation-Based Training on Palliative Caregivers' Hand Hygiene Knowledge and Practices: A Double-Blind Randomized Controlled, Single-Center Study
Brief Title: Handwashing Knowledge and Practice of Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sultanbeyli State Hospital (Other Government)
Responsible Party: Principal Investigator, murat koç, Principal Investigator, Istanbul Sultanbeyli State Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2023s01
Record Dates: First submitted 2023-04-16; First posted 2023-05-08 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hand Hygiene
Keywords: Palliative Care; Hand Hygiene; Simulation Training

STUDY DESIGN:
Intervention Model Description: Preliminary information will be given to the experimental group before the application of the simulation. After the preliminary information, training will be given to the experimental group. In addition, how to provide hand washing will be shown with a demonstration method. After the training, the simulation application will be carried out. After the simulation application is completed, the attendants will be asked to make their self-evaluations. Then, a second feedback will be given by the trainer and the analysis session will be terminated. A handwashing brochure will be provided after the study data has been collected.
  No intervention will be applied to the control group after the pre-test. A handwashing brochure will be provided after the study data has been collected.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand hygiene training (Active Comparator): Hand hygiene theoretical training and simulation application
  Interventions: Other: hand hygiene theoretical + simulation training
- Observation group (Placebo Comparator): Hand hygiene theoretical training was given.
  Interventions: Other: hand hygiene theoretical training

INTERVENTIONS:
Other: hand hygiene theoretical training — Hand hygiene theoretical training
  * Powerpoint presentation,
  * How to ensure hand hygiene according to the demonstration method,
  Arms: Observation group
Other: hand hygiene theoretical + simulation training — Hand hygiene theoretical training
  * Powerpoint presentation,
  * How to ensure hand hygiene according to the demonstration method,
  Hand hygiene simulation training will be carried out by the researcher in an environment with a sink.
  * Simulation-based training on standard patients,
  * Hand hygiene application and important points to be considered during the application will be emphasized.
  Arms: Hand hygiene training

SUMMARY:
This study was planned as a randomized controlled study to evaluate the effect of hand hygiene training given to the companions in the palliative care service with standard patient simulation on hand washing knowledge and practices.

Companions who are over the age of eighteen, who are at least literate, who can communicate effectively, and who fully fill in the data collection tools will be included in the study.

The key questions it aims to answer Does the hand hygiene training given with standard patient simulation have an effect on the hand washing knowledge of the attendants? Do the attendants participating in the hand hygiene training given with standard patient simulation have an effect on hand washing practices?

DETAILED DESCRIPTION:
Palliative care is an interdisciplinary approach that provides health care services for patients with cancer, Alzheimer's, chronic diseases and organ failure such as heart, lung and kidney and provides treatment and support services by including family members in order to reduce pain, manage symptoms and improve quality of life in patients. is the approach.

Palliative care can be provided in hospitals, primary health care institutions, home settings and nursing homes. The economic difficulties of individuals in meeting the health care services offered in hospitals and the difficulties in reaching health care institutions have revealed the necessity of home care services. However, the inability of sick individuals to receive regular and effective home care services by the same health professionals has created different problems. Although palliative care has been established rapidly in our country, the number and training of health professionals is insufficient. Therefore, it becomes difficult to provide services to individuals in need of health care.

Factors such as inadequacies in the management of symptoms in the palliative care process, worsening of the disease prognosis and inability to provide the necessary medical support create many problems.The complexity of palliative care also creates problems in providing quality care to patients. Caregiving is not only limited to helping, but also provides support in terms of physical, mental, psychological, social and economic aspects. Experienced in the maintenance process; The characteristics of the care environment and the insufficient support affect the relatives of the patients negatively.As a result of these situations, the relatives of the patients are involved in a difficult situation to cope with.

Generally, first-degree relatives of the patients undertake the duty of accompanying them. The companion practice, which is accepted among the patient rights, meets the needs of the patients due to the low number of nurses. While the companions experience emotional problems due to their closeness to the sick individuals, they also have auxiliary roles such as helping the patient to eat, making him move, helping him get dressed or dressed, drinking his medication under the control of health professionals, and changing the bed linens.

Palliative care patients are the group most affected by infections due to invasive procedures for diagnosis and treatment, complications, weak immune system of the patient, and existing acute and chronic diseases. One of the most effective and easy ways to control infections and prevent their spread, both in daily life and in hospitals, is to provide hand hygiene. In hospital settings, infection prevention and control procedures recognize hand washing as the primary solution. Poor hand hygiene increases the risk of nosocomial infections, which negatively affect the patient's treatment, cause health complications, and thus prolong the hospital stay. In controlling hospital infections, hand hygiene behaviors and awareness of patient companions, who have an important place in the care of patients, should be considered as well as the hand hygiene behaviors and awareness of healthcare professionals in palliative care. Warning measures such as hand hygiene education related to prevention of nosocomial infections can reduce the risk of transmission. In a study conducted in 2019, it was determined that repeated trainings on hand hygiene and the posters prepared improved the hand hygiene of the companions. In the study conducted in 2015, it was stated that the hand hygiene of health professionals and companions will ensure the prevention and control of infections and that the trainings given will increase their hand hygiene behavior and awareness. In addition, in the study conducted in 2014, in which the hand hygiene compliance of the auxiliary service personnel was investigated, it was determined that education was effective on the hand hygiene compliance of the auxiliary service personnel. İt was determined that the hand hygiene compliance status would develop positively as the information about hand hygiene increased.

While the studies on hand hygiene in the literature deal with healthcare professionals, there is no study on hand hygiene of the companions who support the patient's care in the palliative care process. In order to protect patients from infection in the palliative care process, it is very important to evaluate the companions within the chain of infection and to support them in order to provide appropriate hand hygiene.

The study was planned to evaluate the effect of hand hygiene training given to the companions in the palliative care service with standard patient simulation on hand washing knowledge and practices.

ELIGIBILITY:
Inclusion Criteria:

* Over eighteen years old
* Least literate
* Able to communicate effectively
* Filling the data collection tools completely

Exclusion Criteria:

* Under the age of eighteen
* İlliterate
* No effective communication
* İncomplete data collection tools

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-09-17 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Hand Washing Information Evaluation Form | 4 weeks
  Before starting the research, "Hand Hygiene Practice Inventory", "Hand Hygiene Compliance Scale for auxiliary service personnel", "Social Hand Washing Attitude Scale" and clinical observations were adapted to the palliative care process by the researchers and submitted to the approval of 8 experts. The "Hand Washing Information Evaluation Form", which evaluates the awareness of handwashing and the behavior of the patient about which interventions to apply hand hygiene, consists of 23 questions in total. Participants can get points between 23 and 112. Higher scores indicate better knowledge.
Hand Washing Applications Evaluation Form | 4 weeks
  The "Hand Washing Applications Evaluation Form", which was adapted to the palliative care process by the researchers in line with the World Health Organization's Hand Hygiene Guidelines and submitted to the approval of 8 experts, and which provides control of the handwashing practices of the participants, consists of a total of 18 check-list. Participants can get points between 0 and 18. Higher scores indicate better applications.

CONTACTS AND LOCATIONS:
Locations (1):
- Sultanbeyli Devlet Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allegranzi B, Pittet D. Role of hand hygiene in healthcare-associated infection prevention. J Hosp Infect. 2009 Dec;73(4):305-15. doi: 10.1016/j.jhin.2009.04.019. Epub 2009 Aug 31. PMID 19720430
- [Background] Fox C, Wavra T, Drake DA, Mulligan D, Bennett YP, Nelson C, Kirkwood P, Jones L, Bader MK. Use of a patient hand hygiene protocol to reduce hospital-acquired infections and improve nurses' hand washing. Am J Crit Care. 2015 May;24(3):216-24. doi: 10.4037/ajcc2015898. PMID 25934718
- [Background] Kavalieratos D, Gelfman LP, Tycon LE, Riegel B, Bekelman DB, Ikejiani DZ, Goldstein N, Kimmel SE, Bakitas MA, Arnold RM. Palliative Care in Heart Failure: Rationale, Evidence, and Future Priorities. J Am Coll Cardiol. 2017 Oct 10;70(15):1919-1930. doi: 10.1016/j.jacc.2017.08.036. PMID 28982506
- [Derived] Yalcin Atar N, Koc M. The Effect of Simulation-Based Training on the Hand Hygiene Knowledge and Practices of Palliative Caregivers: A Double-Blind, Randomized, Controlled Single-Center Study. Nurs Health Sci. 2024 Sep;26(3):e13164. doi: 10.1111/nhs.13164. PMID 39301983